CLINICAL TRIAL: NCT06450197
Title: A Double-blind, Placebo-controlled Phase IIa Study to Evaluate the Efficacy and Safety of AZD7798 in Patients With Moderate to Severe Crohn's Disease
Brief Title: Phase IIa Study Evaluating AZD7798 in Crohn's Disease
Acronym: AMALTHEA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9690C00005
Record Dates: First submitted 2024-05-08; First posted 2024-06-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Moderate to Severe Crohn's Disease
Keywords: Crohn disease; Inflammation
MeSH Terms: conditions — Crohn Disease; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD7798 (Experimental): AZD7798
  Interventions: Drug: AZD7798
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD7798 — AZD7798
  Arms: AZD7798
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, parallel group, placebo-controlled Phase IIa study designed to evaluate the efficacy and safety of AZD7798 in participants with moderate to severe Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age.
2. Diagnosis of Crohn's disease established with verifiable clinical, AND at least one of imaging, endoscopic and/or histopathologic evidence.
3. Moderate to severe active Crohn's disease.
4. Ileal/ileocecal (L1), colonic (L2), or ileocolonic (L3) disease, as classified based on the localisation of active inflammation.
5. Capable of giving signed informed consent.
6. A history of at least one of:

   1. Intolerance or inadequate response to conventional treatment (oral corticosteroid, azathioprine, 6-mercaptopurine, or methotrexate), biologics, or other approved advanced therapy (eg, JAK inhibitors) OR
   2. Corticosteroid dependency (defined as inability to taper below budesonide 6 mg/day or prednisolone 10 mg/day equivalent dosing without recurrent active disease) for the treatment of Crohn's disease.

Exclusion Criteria:

1. Evidence, or clinical suspicion, of other forms of IBD or concomitant additional active gastrointestinal luminal inflammatory diseases.
2. Known symptomatic strictures or bowel stenoses or strictures preventing passage of endoscope throughout the colon.
3. Any complications of Crohn's disease where surgery is anticipated or planned prior to end of study treatment.
4. Evidence of extensive prior gastrointestinal surgical interventions.
5. Within 3 months prior to screening endoscopy visit:

   1. History of toxic megacolon
   2. Diagnosis of peritonitis or need for treatment of peritonitis
   3. Bowel perforation or evidence of obstruction.
6. All intrabdominal abscesses are excluded. Cutaneous and perianal/perirectal abscesses and fistulae are excluded unless adequately drained at least 4 weeks prior to screening endoscopy visit with no anticipation for surgery prior to end of study treatment.
7. Ongoing or expected nutritional dependency on total enteral or parenteral nutrition during study.
8. Evidence of an increased risk of colorectal cancer.
9. Symptomatic oral Crohn's disease within one year.
10. Any of the following treatments within the specified time period prior to screening endoscopy visit

    1. An anti-TNF biologic within 8 weeks prior to screening endoscopy visit
    2. Any biologic targeting immune response other than an anti-TNF within 12 weeks prior to screening endoscopy visit
    3. Other advanced small molecule treatments for Crohn's disease within 4 weeks prior to screening endoscopy visit
    4. Cyclosporine, mycophenolate mofetil, sirolimus (rapamycin), thalidomide, or tacrolimus (FK-506) within 4 weeks prior to screening endoscopy visit
    5. Treatment with apheresis within 4 weeks prior to screening endoscopy visit
    6. Administration of any live vaccine within 4 weeks prior to screening endoscopy visit to end of study
    7. Faecal microbiota transplantation within 4 weeks prior to screening endoscopy visit
    8. Lymphocyte-depleting treatment within 12 months prior to screening endoscopy visit
    9. Any previous exposure to AZD7798.
11. Any changes in dosing of the following medications prior to screening endoscopy visit as outlined:

    1. 5-aminosalicylates within 2 weeks
    2. Oral corticosteroids within 2 weeks or stable doses of steroids exceeding the following dose equivalents:

    (i) Systemic steroids > 20 mg/day or prednisolone equivalent (ii) Locally targeted steroids exceeding maximum budesonide dose equivalent (9 mg/day) (c) Immunomodulators within 4 weeks (d) Antibiotic therapy for the treatment of Crohn's disease (e) Probiotics within 2 weeks.
12. Known or suspected history of chronic use of nonsteroidal anti-inflammatory drugs.
13. Evidence of recent or currently active infection, including use of IV or oral antibiotics for documented infection within 30 days prior to screening endoscopy visit.
14. Evidence of chronic HBV or HCV.
15. History of TB (active or latent) unless an appropriate course of treatment has been completed.
16. Positive diagnostic TB test at screening.
17. History of serious opportunistic infection within 12 months prior to screening endoscopy visit.
18. CMV colitis within previous 12 months prior to screening endoscopy visit.
19. Positive C. difficile toxin stool test at screening.
20. Symptomatic herpes zoster infection within 3 months prior to screening endoscopy.
21. Any identified immunodeficiency.
22. Abnormal laboratory results at screening suggesting participation may be unsafe, which will prevent the patient from completing the study, or will interfere with the interpretation of the study results.
23. Reproduction:

    1. Pregnant and breastfeeding patients, or those planning to breastfeed during the study
    2. FOCBP unless completely abstinent or using a highly effective contraception and barrier method of contraception.
24. Prolonged QTcF interval.
25. Clinically significant cardiovascular conditions.
26. Current malignancy or history of malignancy.
27. Current significant major or unstable respiratory disease, heart disease, cerebrovascular disease, haematological disease, hepatic disease, renal disease, gastrointestinal disease or other major disease other than active Crohn's disease.
28. Current enrolment in another interventional study or treatment with any investigational drug within 4 months prior to screening endoscopy visit.
29. Unstable lifestyle factors.
30. Patients committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
31. Investigator concerns regarding patient's willingness and ability to attend all study visits, comply with the study procedures, read in order to complete questionnaires, or to complete the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
CDAI remission | Week 12
  Crohn's Disease Activity Index (CDAI) is a research tool used to quantify the symptoms of patients with Crohn's disease. It is based on: number of loose stools, abdominal pain, general well-being, extraintestinal complications, antidiarrheal agents used in the previous 7 days, abdominal mass felt on palpation, hematocrit and body weight

SECONDARY OUTCOMES:
Endoscopic response | Week 12
  Simple Endoscopic Score for Crohn's Disease (SES-CD) is based on the evaluation of five defined bowel segments (rectum, sigmoid + descending colon, transverse colon, ascending colon, and terminal ileum), and in these segments the presence and size of ulcerations and the extent of the inflammatory area and stenosis are assessed
Endoscopic remission | Week 12
  Simple Endoscopic Score for Crohn's Disease (SES-CD) is based on the evaluation of five defined bowel segments (rectum, sigmoid + descending colon, transverse colon, ascending colon, and terminal ileum), and in these segments the presence and size of ulcerations and the extent of the inflammatory area and stenosis are assessed
Endoscopic score change from baseline | Week 12
  Simple Endoscopic Score for Crohn's Disease (SES-CD) is based on the evaluation of five defined bowel segments (rectum, sigmoid + descending colon, transverse colon, ascending colon, and terminal ileum), and in these segments the presence and size of ulcerations and the extent of the inflammatory area and stenosis are assessed
CDAI response | Week 12
  Crohn's Disease Activity Index (CDAI) is a research tool used to quantify the symptoms of patients with Crohn's disease. It is based on: number of loose stools, abdominal pain, general well-being, extraintestinal complications, antidiarrheal agents used in the previous 7 days, abdominal mass felt on palpation, hematocrit and body weight
CDAI score change from baseline | Week 12
  Crohn's Disease Activity Index (CDAI) is a research tool used to quantify the symptoms of patients with Crohn's disease. It is based on: number of loose stools, abdominal pain, general well-being, extraintestinal complications, antidiarrheal agents used in the previous 7 days, abdominal mass felt on palpation, hematocrit and body weight
Symptomatic remission | Week 12
  Decrease of average daily stool frequency and average daily abdominal pain
Serum AZD7798 concentration | Up to 85 days
  Serum AZD7798 concentration (PK)
Incidence of anti-drug antibody response | Up to 36 weeks
  Incidence of anti-drug antibody (ADA) response - number and percentages with a positive ADA result
Titre of anti-drug antibody response | Up to 36 weeks
  Titre of anti-drug antibody (ADA) response - immunogenicity titre will be summarized descriptively as a continuous variable, only for ADA positive tests

CONTACTS AND LOCATIONS:
Locations (168):
- United States (23):
  - Research Site, Phoenix, Arizona
  - Research Site, Escondido, California
  - Research Site, La Jolla, California
  - Research Site, Victorville, California
  - Research Site, Hamden, Connecticut
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Idaho Falls, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, Ann Arbor, Michigan
  - Research Site, Clinton Township, Michigan
  - Research Site, Liberty, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Uniontown, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Garland, Texas
  - Research Site, Mansfield, Texas
  - Research Site, San Antonio, Texas
- Argentina (6):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad Autonoma de Bs As
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Quilmes
  - Research Site, San Miguel de Tucumán
- Australia (11):
  - Research Site, Adelaide
  - Research Site, Bedford Park
  - Research Site, Box Hill
  - Research Site, Epping
  - Research Site, Fitzroy
  - Research Site, Heidelberg
  - Research Site, Liverpool
  - Research Site, Melbourne
  - Research Site, Parkville
  - Research Site, South Brisbane
  - Research Site, Wollongong
- Austria (2):
  - Research Site, Klagenfurt
  - Research Site, Vienna
- Belgium (4):
  - Research Site, Aalst
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (7):
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Jaú
  - Research Site, Porto Alegre
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (3):
  - Research Site, Gorna Oryahovitsa
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (2):
  - Research Site, Lethbridge, Alberta
  - Research Site, Vaughan, Ontario
- Chile (3):
  - Research Site, Santiago
  - Research Site, Talcahuano
  - Research Site, Viña del Mar
- China (7):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Wuhan
- Croatia (3):
  - Research Site, Osijek
  - Research Site, Rijeka
  - Research Site, Zagreb
- France (5):
  - Research Site, Amiens
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Pierre-Bénite
  - Research Site, Vandœuvre-lès-Nancy
- Germany (7):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Halle
  - Research Site, Jena
  - Research Site, Kiel
  - Research Site, Potsdam
  - Research Site, Ulm
- Hungary (3):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Gyöngyös
- Italy (4):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Roma
  - Research Site, Rome
- Japan (17):
  - Research Site, Asahikawa-shi
  - Research Site, Chiba
  - Research Site, Hamamatsu
  - Research Site, Hirosaki-shi
  - Research Site, Hiroshima
  - Research Site, Kamakura-shi
  - Research Site, Kashiwa-shi
  - Research Site, Kure-shi
  - Research Site, Minatoku
  - Research Site, Morioka
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Sakura-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
- Malaysia (5):
  - Research Site, Johor Bahru
  - Research Site, Kota Bharu
  - Research Site, Kota Kinabalu
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
- Mexico (6):
  - Research Site, Durango
  - Research Site, Mexico City
  - Research Site, Mérida
  - Research Site, México
  - Research Site, Tlajomulco de Zúñiga
  - Research Site, Veracruz
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Nijmegen
  - Research Site, Tilburg
- Poland (8):
  - Research Site, Bydgoszcz
  - Research Site, Chojnice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Sopot
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Timișoara
- Slovakia (4):
  - Research Site, Košice
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Trnava
- South Africa (4):
  - Research Site, Assagay
  - Research Site, Cape Town
  - Research Site, Milnerton
  - Research Site, Plumstead
- Spain (5):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Seville
- Sweden (2):
  - Research Site, Linköping
  - Research Site, Stockholm
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (7):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, İzmit
  - Research Site, Malatya
- Ukraine (5):
  - Research Site, Chernivtsі
  - Research Site, Kiev
  - Research Site, Kyiv
  - Research Site, Ternopil
  - Research Site, Vinnytsia
- Vietnam (4):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Hồ Chí Minh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/